CLINICAL TRIAL: NCT03649815
Title: Testing the Feasibility and Outcomes of a Digital Health Support for Individuals With Schizophrenia Spectrum Mental Illnesses
Brief Title: Feasibility and Outcomes of a Digital Health Support for the Schizophrenia Spectrum
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Sean Kidd, Senior Scientist, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 84-2016
Record Dates: First submitted 2018-08-23; First posted 2018-08-28 (Actual); Results first posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Schizophrenia Spectrum and Other Psychotic Disorders
Keywords: schizophrenia; psychosis; mHealth; digital health
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders; Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Use of mHealth Technology (Experimental): This single arm of the study involves the provision of the mobile health technology entitled App4Independence.
  Interventions: Combination Product: App4Independence

INTERVENTIONS:
Combination Product: App4Independence — The mobile, app-based platform was designed to:
  * Help prevent social isolation through personalized prompts, scheduling of activities, and connections to a range of resources relevant to social engagement
  * Enhance hopeful and informed engagement in the recovery process through functions that foster resilience and draw on evidence based strategies to enhance wellness (e.g., personalized affirmations; tip sheets; relaxation exercises)
  * Encourage and check-in on daily essential activities for patients - addressing memory, attention, and initiation challenges that often occur as a part of this illness
  * Provide basic health/safety functionality and track level of wellness
  * Provide an anonymous peer-peer online network for strategy sharing
  * Provide an ambient sound detector to assist with identifying hallucinations

SUMMARY:
This protocol describes an attempt to capture the development phase of a mobile support for individuals with schizophrenia. The intent is to describe and account for a rigorous development process that will result in the creation of a beta version that would be tested in a randomized trial for effectiveness - to be addressed in a subsequent protocol

DETAILED DESCRIPTION:
General Issues The most common contributors to relapse in schizophrenia and associated mental illnesses are medication non-adherence, social isolation, and inadequate supports. Driven to a large extent by system of care shortcomings and the many challenges presented by symptoms, the impacts of these problems are profound from individual to system levels. This is a global issue, and to date technology has not been substantively leveraged in generating solutions - despite evidence of substantial uptake of relevant technologies by relevant populations. To date, there are few products on the market that address the constellation of issues outlined above. It is an area where a nuanced approach is needed as this illness is highly diverse in presentation, attended by a number of social determinants of health that greatly affect outcomes and, quite commonly, ambivalence with respect to service provider and caregiver engagement. This scenario as it exists for schizophrenia stands in sharp contrast with the many thousands of applications developed for other mental health issues.

Cellphone Based Technologies and Schizophrenia There is a small, emergent literature that is examining the feasibility and outcomes of mobile applications that address schizophrenia. Broadly, targeted mobile and online applications in areas such as cognitive remediation (brain training games) have been found feasible and do not result in any noted risks in their use and there have been promising findings in outcome studies of emergent mHealth strategies for schizophrenia of the kind tested here.

Local Work in this Area to Date

Initial mapping of key domains relevant to an app in this area has been conducted based upon the experience of the collaborators and an understanding of the relevant practice literatures. This initial draft, which might be considered a 'paper prototype', let to the identification of the following needs:

The platform would:

* Help prevent social isolation through personalized prompts, scheduling of activities, and connections to a range of resources relevant to social engagement
* Enhance hopeful and informed engagement in the recovery process through functions that foster resilience and draw upon evidence based strategies to enhance wellness (e.g., personalized affirmations; tip sheets; relaxation exercises)
* Facilitate automated support and link to caregivers
* Encourage and check-in on daily essential activities for patients - addressing memory, attention, and initiation challenges that often occur as a part of this illness
* Provide basic health/safety functionality and track level of wellness

Specifically, the app was designed to be made up of 4 functional areas:

1. A needs assessment in order to determine care/interaction pathway, crisis planning and routine builders, accompanied by ongoing assessment to keep components relevant and engaging and to facilitate treatment planning and support by providers.
2. Daily interactions and check-in functionality for self-determination of messaging, reward messaging, social interaction content.
3. An algorithm to determine content based on ambient and interaction data content triggers and risk flagging built on evidence-based guidelines.
4. Self-Management portal and caregiver dashboard.

Research Objective

This study was undertaken to engage in a rigorous process of feasibility testing. This will then be followed by a randomized trial of the beta version that will be generated through the process outlined in this protocol (will be the subject of a subsequent protocol and not addressed here). As such, the objective of this research is to capture and record the process of development of a functional, beta version of this technology. This test includes outcome data derived from 1 month of app use comprised of both qualitative feedback and quantitative outcome data. The objective is to determine feasibility prior to further trials and validation efforts.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 years of age or older
* Have a schizophrenia spectrum diagnosis
* Own and regularly use a smart phone equipped with an Android operating system and a talk and data plan
* Read and speak conversational English

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2018-05-08 (Actual); Study Completion 2018-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean Kidd, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available via a supplementary file in the publication.
Supporting Information: Study Protocol
Time Frame: Available upon publication indefinitely.
Access Criteria: Publically accessible.

RESULTS

PARTICIPANT FLOW:
Groups:
- Use of mHealth Technology: This single arm of the study involves the provision of the mobile health technology entitled App4Independence.
  App4Independence: The mobile, app-based platform was designed to:
  * Help prevent social isolation through personalized prompts, scheduling of activities, and connections to a range of resources relevant to social engagement
  * Enhance hopeful and informed engagement in the recovery process through functions that foster resilience and draw on evidence based strategies to enhance wellness (e.g., personalized affirmations; tip sheets; relaxation exercises)
  * Encourage and check-in on daily essential activities for patients - addressing memory, attention, and initiation challenges that often occur as a part of this illness
  * Provide basic health/safety functionality and track level of wellness
  * Provide an anonymous peer-peer online network for strategy sharing
  * Provide an ambient sound detector to assist with identifying hallucinations
Period: Overall Study
Arm/Group | Use of mHealth Technology
Started | 38
Completed | 38
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Use of mHealth Technology
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.42 (8.60)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Transgender | 1
  Male | 27
  Female | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 16
  Black Canadian or African or African Caribbean | 9
  Mixed | 9
  Other | 4
Level of Education [Count of Participants; unit: Participants]
  Junior High/Middle School | 4
  High School | 6
  Tertiary Education | 28
Employment [Count of Participants; unit: Participants]
  Full Time | 2
  Part Time | 6
  Casual | 4
  Student | 11
  Unemployed | 9
  Not In Labour Force | 6
Diagnosis [Count of Participants; unit: Participants]
  Schizophrenia | 24
  Schizoaffective | 9
  Psychosis NOS or Psychosis comorbid with BPD | 1
  ASD with prominent psychosis symptomatology | 1
Age of first illness onsent/Age at 1st Hospitalization [Mean (Standard Deviation); unit: years] | 24.16 (7.70)
Mobile technology use [Count of Participants; unit: Participants]
  Hourly Use | 30
  Daily Use | 8
  Texting (1-5 times/day) | 20
  Emailing (1-5 times/day) | 21
  Social Media (1-5 times/day) | 16
Brief Symptom Inventory [Mean (Standard Deviation); unit: units on a scale] — The Brief Symptom Inventory (BSI) assesses the level of psychiatric symptomatology providing both total and subscale scores. All 53 items are 5-point likert with higher scores meaning higher symptomatology. Overall total can range from 0-212 (average of the subscale totals plus 4 items). Lowest scores for all are 0, with 20 the highest score for hostility, phobic anxiety, paranoid ideation, psychoticism; 16 the highest score for interpersonal sensitivity; 24 the highest for obsessive compulsive, depression, anxiety; and 28 for somatization.Subscale items are averaged to get the subscale total.
  units on a scale
    Total | 46.21 (32.86)
    Psychoticism | 5.34 (4.63)
    Somatization | 4.95 (4.40)
    Depression | 6.47 (5.59)
    Hostility | 2.42 (2.41)
    Phobic Anxiety | 3.90 (4.11)
    OCD | 8.21 (5.06)
    Anxiety | 4.92 (5.50)
    Paranoid Ideation | 4.97 (4.54)
    Interpersonal Sensitivity | 4.45 (3.90)
Personal Recovery Outcome Measure [Mean (Standard Deviation); unit: units on a scale] — Personal Recovery Outcome Measure (PROM) was used to assess degree of engagement in the recovery process. The prom has 30 items, all 5 point likert with higher scores meaning more recovery engagement. The metric is the total score (0-120)/4 to provide an adjusted score. There are no subscales.
  units on a scale | 7.13 (1.66)
Brief Adherence Rating Scale [Mean (Standard Deviation); unit: units on a scale] — Brief Adherence Rating Scale (BARS) was used to examine implications of A4i for medication use. A total score ranging from 0-100 is provided with 100 indicating better adherence.
  units on a scale | 98.27 (3.10)
Living Circumstances [Count of Participants; unit: Participants]
  Alone in private dwelling | 13
  Private dwelling with parents | 9
  With roomates | 9

OUTCOME MEASURES:

1. Primary Outcome: Symptomatology
Description: The Brief Symptom Inventory (BSI) assesses the level of psychiatric symptomatology providing both total and subscale scores. All 53 items are 5-point likert with higher scores meaning higher symptomatology. For the overall score the total is used and can range from 0-212. Total scores from each of the 9 subscales are similarly used with higher scores meaning greater subscale symptomatology. Lowest scores for all are 0, with 20 the highest score for hostility, phobic anxiety, paranoid ideation, psychoticism; 16 the highest score for interpersonal sensitivity; 24 the highest for obsessive compulsive, depression, anxiety; and 28 for somatization.
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Use of mHealth Technology
Number analyzed (Participants) | 38
score on a scale
  Total | 41.66 (33.80)
  Psychoticism | 4.34 (4.23)
  Somatization | 4.29 (5.40)
  Depression | 4.29 (4.57)
  Hostility | 1.97 (2.58)
  Phobic Anxiety | 2.97 (3.75)
  OCD | 6.37 (4.70)
  Anxiety | 4.63 (4.81)
  Paranoid Ideation | 3.71 (3.49)
  Interpersonal Sensitivity | 3.74 (3.94)
Statistical Analysis 1: Comparison: Use of mHealth Technology; Test type: Other; p = 0.067, Paired Sample T-Test
Statistical Analysis 2: Comparison: Use of mHealth Technology; Test type: Other; p = 0.071, Paired Sample T-Test — Controlled for gender, age, and baseline symptomatology

2. Primary Outcome: Recovery Process Engagement
Description: Personal Recovery Outcome Measure (PROM) was used to assess degree of engagement in the recovery process. The prom has 30 items, all 5 point likert with higher scores meaning more recovery engagement. The metric is the total score (0-120)/4 to provide an adjusted score. There are no subscales.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Use of mHealth Technology
Number analyzed (Participants) | 38
score on a scale | 7.45 (1.63)
Statistical Analysis 1: Comparison: Use of mHealth Technology; Test type: Other; p = 0.047, Paired Sample T-Test
Statistical Analysis 2: Comparison: Use of mHealth Technology; Test type: Other; p = 0.036, Paired Sample T-Test — Controlled for gender, age and baseline symptomatology

3. Primary Outcome: Treatment Adherence
Description: Brief Adherence Rating Scale (BARS) was used to examine implications of A4i for medication use. A total score ranging from 0-100 is provided with 100 indicating better adherence.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Use of mHealth Technology
Number analyzed (Participants) | 38
score on a scale | 98.94 (2.35)
Statistical Analysis 1: Comparison: Use of mHealth Technology; Test type: Other; p = 0.032, Paired Sample T-Test
Statistical Analysis 2: Comparison: Use of mHealth Technology; Test type: Other; p = 0.006, Paired Sample T-Test — Controlled for gender, age and baseline symptomatology

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Use of mHealth Technology
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 0/38

LIMITATIONS AND CAVEATS:
No control condition limits comments on effectiveness and ability to control for confounders. The time period might speak to a lack of signal in medication adherence. Cannot speak to how well A4i would perform outside of the research context.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-10-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT03649815/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-05): https://cdn.clinicaltrials.gov/large-docs/15/NCT03649815/ICF_001.pdf